CLINICAL TRIAL: NCT04535726
Title: The Relationship Between Blood Pressure and Arterial Stiffness in HFpEF Patients With Different Levels of Obesity
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Clinical Professor, Chongqing Medical University
Other Study IDs: 2020-08
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: obesity; the level of blood pressure; arterial stiffness
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) was considered as a heterogeneous disease with multi-organ and multi-system design, which is related to various complications, such as hypertension, obesity and arteriosclerosis. Studies have found that hypertension and obesity are respectively associated with increased arterial stiffness. However, there is still no research investigating the the relationship between blood pressure and arterial stiffness in HFpEF patients with different levels of obesity.

DETAILED DESCRIPTION:
Before the 21st century, Heart failure with preserved ejection fraction (HFpEF) was considered as a disease with simple diastolic dysfunction, but after the 21st century, HFpEF was considered as a heterogeneous disease with multi-organ and multi-system design, which is related to various complications, such as hypertension, obesity and arteriosclerosis. Other studies have found that hypertension and obesity are respectively associated with increased arterial stiffness. However, there is still no research investigating the the relationship between blood pressure and arterial stiffness in HFpEF patients with different levels of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged >=18years old;
* Diagnosed with HFpEF.

Diagnostic criteria including:

1. left ventricular ejection fraction ≥50%；
2. with the symptoms and/or signs of heart failure；
3. BNP≥35 pg/mL and/or NTproBNP≥125 pg/mL；
4. at least one additional criterion: relevant structural heart disease(LVH and/or LAE) or diastolic dysfunction

Exclusion Criteria:

* LVEF less than 45% at any time;
* Severe liver failure;
* Other causes of shortness of breath, such as severe pulmonary disease or severe chronic obstructive pulmonary disease;
* Primary pulmonary hypertension;
* Severe valvular disease of the left heart;
* Chronically bedridden or incapacitated;
* Age <18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with preserved ejection fraction (HFpEF)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness | On admission
  The arterial stiffness of HFpEF patients, for example brachial ankle pulse wave velocity, ardioankle vascular index and so on.
The level of blood pressure | On admission
  The level of systolic and diastolic blood pressure of heart failure patients with preserved ejection fraction.

SECONDARY OUTCOMES:
The change from baseline in quality of life | 6 months
  Measured by Minnesota living with heart failure questionnaire. The score ranges from 0 to 105. The higher score means the worse health-related quality of life.
The re-hospitalization rate of heart failure | 6 months
  The re-hospitalization rate of heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, doctor, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun M, Gao L, Bai H, Hu W, Zhang X, Xiao J, Deng X, Tao H, Ge P, Qin Y, Zhang D. Association Between Visceral Fat, Blood Pressure and Arterial Stiffness in Patients with HFpEF: A Mediation Analysis. Diabetes Metab Syndr Obes. 2023 Mar 8;16:653-662. doi: 10.2147/DMSO.S399928. eCollection 2023. PMID 36923684